CLINICAL TRIAL: NCT03003637
Title: ImmunoModulation by the Combination of Ipilimumab and Nivolumab Neoadjuvant to Surgery In Advanced Or Recurrent Head and Neck Carcinoma. Subtitle: Hypoxia as a Determinant for the Effect of Nivolumab With or Without Ipilimumab on Intra-tumoral T Cell Capacity
Brief Title: ImmunoModulation by the Combination of Ipilimumab and Nivolumab Neoadjuvant to Surgery In Advanced or Recurrent Head and Neck Carcinoma
Acronym: IMCISION
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N16IMC
Record Dates: First submitted 2016-12-22; First posted 2016-12-28 (Estimated); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Immunotherapy; Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab with or without Ipilimumab (Experimental): First dose scheme will be 2x nivolumab 240 mg flat dose, weeks 1 and 3. When feasible and safe, the next patients will be treated with the following dose scheme: the combination of 1x ipilimumab 1 mg/kg + nivolumab 240 mg flat dose in week 1 and nivolumab mono-therapy 240 mg flat dose in week 3
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab (240 mg flat dose, week 1 and week 3, twice in total) monotherapy, neoadjuvant to SOC (surgery with or without adjuvant (C)RT).
  Other Names: Nivolumab (Opdivo) BMS-936558-01
Drug: Ipilimumab — Ipilimumab (1 mg/kg) only in week 1, in combination with nivolumab (240 mg flat dose, week 1 and week 3, twice in total), neoadjuvant to SOC (surgery with or without adjuvant (C)RT).
  Other Names: Ipilimumab (Yervoy) BMS

SUMMARY:
This is a phase IB/II trial to examine feasibility and safety of checkpoint blockade (aPD1 with or without aCTLA4) neoadjuvant to standard of care (SOC) in advanced stage head and neck squamous cell carcinoma (HNSCC), a patient population in need for improved clinical outcome and in tumors likely to respond to neoadjuvant aPD1 and aCTLA4. In addition, with this research protocol the potential impact of intratumoral hypoxia on tumor infiltrating lymphocyte (TIL) abundance, differentiation and effector function will be assessed, and the potentially divergent effects of T cell checkpoint blockade in areas of hypoxia and normoxia.

DETAILED DESCRIPTION:
The phase Ib is designed as 3 + 3, with primary objective feasibility and toxicity.

Of Note: endpoints must be reached in all 6 patients of cohort 1 and 2, before start of the next cohort.

The phase II is designed as a single arm design with primary endpoint efficacy.

In phase Ib, two cohorts will be used (cohort 1: nivolumab only and cohort 2: nivolumab and ipilimumab neoadjuvant to surgery) to define which neoadjuvant immunotherapy regimen will be taken towards the expansion cohort 3.

Thirty-two patients will be treated with nivolumab (240 mg flat dose, week 1 and week 3, twice in total) as a single agent OR the combination of ipilimumab (1 mg/kg) + nivolumab (240mg flat dose) in week 1, and nivolumab 240mg flat dose in week 3, neoadjuvant to SOC (surgery with or without adjuvant (C)RT).

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 years and older
* Patients with histologically confirmed T3-4N0-3M0 HNSCC (with soft tissue infiltration depth of ≥ 1 cm) of the oral cavity, oropharynx, hypopharynx or supraglottic larynx, eligible for curative surgery as primary treatment or salvage surgery after failed (chemo)radiation.
* Performance Status ECOG 0 or 1
* No immunosuppressive medications within 6 months prior study inclusion
* Screening laboratory values must meet the following criteria: WBC ≥ 2.0x109/L, Neutrophils ≥ 1.5x109/L, Platelets ≥ 100 x109/L, Hemoglobin ≥ 5.5 mmol/L, Creatinine ≤ 1.5x ULN, AST ≤ 3 x ULN, ALT ≤ 3 x ULN, Total Bilirubin ≤1.5 X ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
* No hard-drug abuse.
* Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives after the last dose of investigational drug.
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of nivolumab w/wo ipilimumab.
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year Men receiving nivolumab w/wo ipilimumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product.
* Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) as well as azoospermic men do not require contraception.
* All subjects must have signed and dated the written informed consent.

Exclusion Criteria:

* Distant metastasis
* Active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical corticosteroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Prior systemic treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways;
* Patients will be excluded if they are positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection;
* Patients will be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS);
* Allergies and Adverse Drug Reaction: history of allergy to study drug components, history of severe hypersensitivity reaction to any monoclonal antibody.
* Underlying medical conditions that, in the Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity determination or adverse events;
* Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids;
* Use of other investigational drugs before study drug administration 30 days and 5 half times before study inclusion;
* Pregnant or nursing.
* As there is potential for hepatic toxicity with nivolumab or nivolumab/ipilimumab combinations, drugs with a predisposition to hepatotoxicity should be used with caution in patients treated with nivolumab-containing regimen.
* In those patients who have a contraindication for cisplatin chemotherapy, Cetuximab might be used as a radiosensitizer for radiotherapy if adjuvant treatment is deemed necessary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2019-10-12 (Actual); Study Completion 2021-02-12 (Actual)

PRIMARY OUTCOMES:
Phase Ib: the number of patients that will not endure a delay in surgery due to neoadjuvant immunotherapy related toxicity OR toxicity due to the treatment of immunotherapy related toxicity. | 2.5 years
Phase II: Tumor response to neoadjuvant IT in terms of tumor tissue pathological response at time of surgery compared to RECIST 1.1 (FDG-PET and perfusion and diffusion weighted MRI). | 2.5 years
Phase Ib/II: the potential impact of local tumor hypoxia on tumor T-cell abundance and capacity before and after neo-adjuvant immunotherapy, through HX4-PET-guided tumor biopsies from hypoxic and normoxic tumor regions. | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lotje Zuur, MD, PhD, Principal Investigator — NKI-AvL
Locations (1):
- NKI-AVL, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vos JL, Zuur CL, Smit LA, de Boer JP, Al-Mamgani A, van den Brekel MWM, Haanen JBAG, Vogel WV. [18F]FDG-PET accurately identifies pathological response early upon neoadjuvant immune checkpoint blockade in head and neck squamous cell carcinoma. Eur J Nucl Med Mol Imaging. 2022 May;49(6):2010-2022. doi: 10.1007/s00259-021-05610-x. Epub 2021 Dec 27. PMID 34957526
- [Derived] Vos JL, Elbers JBW, Krijgsman O, Traets JJH, Qiao X, van der Leun AM, Lubeck Y, Seignette IM, Smit LA, Willems SM, van den Brekel MWM, Dirven R, Baris Karakullukcu M, Karssemakers L, Klop WMC, Lohuis PJFM, Schreuder WH, Smeele LE, van der Velden LA, Bing Tan I, Onderwater S, Jasperse B, Vogel WV, Al-Mamgani A, Keijser A, van der Noort V, Broeks A, Hooijberg E, Peeper DS, Schumacher TN, Blank CU, de Boer JP, Haanen JBAG, Zuur CL. Neoadjuvant immunotherapy with nivolumab and ipilimumab induces major pathological responses in patients with head and neck squamous cell carcinoma. Nat Commun. 2021 Dec 22;12(1):7348. doi: 10.1038/s41467-021-26472-9. PMID 34937871